CLINICAL TRIAL: NCT06872775
Title: A Multi-Center Observational Study to Validate RNA-Biomarkers as Prognostic of Fracture Healing
Brief Title: 855303-RNA Biomarker Validation
Acronym: 855303-RNAVal
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: PharPoint Research, Inc. (Industry); Children's Hospital of Philadelphia (Other); Cooperative Human Tissue Network - Eastern Division (CHTN-ED) (Unknown); Osetomics, LLC (Unknown); Resonant Clinical/Therapak, Claremont, California (Unknown); ResearchDx, Irvine, CA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 855303; UPCC-02924 (Other: University of Pennsylvania Cancer Center (UPCC)); 50526 (Other: SMART IRB)
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fractures, Bone
Keywords: Traumatic Fracture; Appendicular skeleton; long bone; Normal healing; delayed healing; nonunion or non-union or non union; peripheral blood; prognosis
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood will be collected into PAXgene Blood RNA Tubes which protect and stabilize RNA but not other molecules like DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New Traumatic Fractures: Anyone age 18 or over presenting to participating sites for care of new, traumatic appendicular fractures.
  Interventions: Other: Blood draws to assess RNA expression levels

INTERVENTIONS:
Other: Blood draws to assess RNA expression levels — None. Standard of Care (SOC) only.

SUMMARY:
The purpose of this study is to test the accuracy of using RNA in blood as a way to forecast new fracture healing outcome.

DETAILED DESCRIPTION:
This study will follow a registry + biospecimen collection format. Subjects will be enrolled at participating Sites as they present for care for new traumatic appendicular skeletal fractures (0 - ≤7 Days post-injury) and will provide blood specimens for study analysis and future use at up to 4 post-injury windows of treatment (i.e., Window 1, 0 - ≤7 Days; Window 2, 8 - ≤14 days; Window 3, 15 - ≤42 Days; and Window 4, 43 - ≤84 Days post-injury).

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a potential subject must meet ALL of the following criteria:

1. Provision of informed consent for study participation for self in the English language as indicated by a signed and dated, current, and IRB-approved Informed Consent Form (ICF) from

   1. patients making their own SOC clinical decisions prior to the time of the 1st blood sample collection, or
   2. persons initially unable to make their own SOC clinical decisions, who regain capacity to make clinical care decisions after study blood sample collection during the enrollment window and/or before hospital discharge.
2. Patient is expected to receive follow-up SOC fracture care at the Site.
3. Either biological sex at birth (i.e., male or female).
4. Any self-determined gender or sexual preference.
5. Any race and/or ethnicity combination.
6. Age 18 years or older at the time of enrollment; no maximum age.
7. Body weight estimated to be or measured at ≥110 lbs.
8. Presentation for care within 7 calendar days of injury for at least one new traumatic fracture of any bone in the appendicular skeleton with or without additional fractures of the appendicular or axial skeleton and with or without any other traumatic injuries.

   1. A qualifying fracture:

      * May be open or closed as locally defined per SOC.
      * May be displaced or non-displaced per SOC.
      * Must result from blunt or penetrating trauma.
      * May not be in a location of the body that was chronically paralyzed pre-trauma or has become permanently paralyzed because of the trauma.
      * Does not include traumatic amputation above the fracture Site for qualifying fractures
   2. Index treatment plan:

      * May be operative or non-operative.
      * May include staged treatment with or without the use of external fixators, and/or antibiotic beads, and/or other planned intervention.
      * Does not include hemi- or total arthroplasty to treat the qualifying fracture.
      * Does not include amputation above the qualifying fracture.
9. In good general health as evidenced by clinical presentation and/or medical history and without any diagnoses that preclude a life expectancy of at least 2 years after injury.
10. No healed or unhealed fractures within 12 months prior to the event resulting in the qualifying fracture.
11. Blood collection through venipuncture at the volume and frequency per protocol is not contraindicated either through past medical history or current clinical status
12. 45 CFR 46 Subpart B: For females of reproductive potential: not pregnant at the time of study enrollment.
13. CFR 46 Subpart C: Does not meet the CFR definition of Prisoner.
14. Other vulnerable populations:

    1. Not an individual with pre-existing or newly acquired permanently impaired decision-making capacity , and/or
    2. Not an individual who would be considered an economically or educationally disadvantaged person prior to the qualifying injury as determined by the Site study team per Site standards.

       -

Exclusion Criteria

An individual who meets ANY of the following criteria will be excluded from participation in this study:

1. Enrolled in another research study that requires any study-specific blood draws from 0 - ≤84 Days post-injury or a study that prohibits co-enrollment of any kind.
2. Traumatic injuries at presentation are limited to soft tissue injuries and/or axial skeletal fractures.
3. The presentation appendicular fractures is a result of pathological not traumatic mechanism
4. Any other circumstances that in the opinion of the PI would either put the successful completion of the study at risk, and/or which makes study participation unduly burdensome to the Subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who provide blood samples and whose clinically determined fracture outcome is known.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-08-24 (Estimated); Study Completion 2028-08-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with correct predicted outcome | 0 - 270 days
  The proportion of Subjects who have a correctly prognosed Fracture Healing Outcome (Normal Healing vs. Delayed Healing vs Nonunion) via RNA in peripheral blood when captured during four specific Windows:
  1. 0 - ≤7 Days post-injury; and/or
  2. 8 - ≤14 days post-injury; and/or
  3. 15 - ≤42 Days post-injury; and/or
  4. 43 - ≤84 Days post-injury
  as compared to clinically determined outcomes up to 270 Days post-injury.
Intra-Patient Correlation | 0 - 270 days
  The intra-patient correlation of RNA-biomarker-driven prognostic calls made by the blinded statistician across windows for those patients who contribute >1 specimen for RNA-biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Mehta, MD, Principal Investigator — University of Pennsylvania; Annamarie D Horan, MPA, PhD, Study Director — University of Pennsylvania
Locations (7):
- United States (7):
  - University of California, Davis Medical Center, Sacramento, California
  - Indiana University, Bloomington, Indiana
  - University of Missouri, Columbia, Missouri
  - Wake Forest University Health Sciences/Advocate Health, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided